CLINICAL TRIAL: NCT02682524
Title: Phase IV Clinical Trial to Evaluate the Efficacy and Safety of PlbCR and Aceclofenac in the Treatment of Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW_PlbCR_401
Record Dates: First submitted 2015-10-12; First posted 2016-02-15 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — aceclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- test (Active Comparator)
  Interventions: Drug: Pelubiprofen CR 45mg tab.
- reference (Active Comparator)
  Interventions: Drug: Aceclofenac 100mg tab.

INTERVENTIONS:
Drug: Pelubiprofen CR 45mg tab.
  Arms: test
Drug: Aceclofenac 100mg tab.
  Arms: reference

SUMMARY:
A multicenter, randomized, double-blinded, parallel, active-controlled, phase IV clinical trial to evaluate the efficacy and safety of PlbCR and aceclofenac in the treatment of patients with osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

* both male and female who is over 35year-old and below 80year-old
* patient who diagnosed as Kellgren & Lawrence stage I~III by X-ray
* osteoarthritis patient who is stable within 3months form starting this clinical trial
* patient who is over 40mm in 100mm Pain VAS at Visit 2
* patient who agreed to participate this clinical trial spontaneously

Exclusion Criteria:

* second osteoarthritis
* patient who has inflammatory disease which can effect efficacy outcomes such as bursitis, tenosynovitis, rheumatoid arthritis, etc.
* patient who diagnosed as gastric ulcer or GI disease by esophagogastroduodenoscopy
* patient who had joint surgery within 12months form screening visit of this clinical trial or planned to operate in this clinical trial period
* patient who has had artificial joint surgery of knee
* malignant tumor patient
* patient who has taken Psychopharmaceutical or Narcotic Analgesics over 3months continuously
* patient who took steroid by oral, inhalation or intraarticular injection within 3months form screening visit of this clinical trial
* patient who took intraarticular hyaluronic acid injection of knee within 2months form screening visit of this clinical trial
* patient who cannot take NSAIDs because of disease or medicine
* allergy of aspirin of other NSAIDs
* patient who has to handle his/her pain by or for CABG
* galactose intolerance, Lactose Intolerance or glucose-galactose malabsorption
* inflammatory bowel disease such as ulcerative colitis or Crohn's disease
* moderate renal disease
* moderate hepatic disease
* moderate hypertension(SBP=>160mmHg, DBP=>100mmHg)
* female who consents to contracept
* patient who is not appropriate for this clinical trial

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline 100mm Pain VAS at 4weeks | 4weeks

SECONDARY OUTCOMES:
Change from baseline 100mm Pain VAS at 2weeks | 2weeks
Change from baseline K-WOMAC Scale at 2weeks and 4weeks | 2weeks, 4weeks
Patient Global Assessment | 4weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Inha university hospital, Chung Gu, Incheon, South Korea